CLINICAL TRIAL: NCT04897854
Title: TIming of Start of systemIc Treatment for Asymptomatic MEtastasized PANcreatic Cancer (TIMEPAN): a Randomized Controlled Multicenter Trial
Brief Title: Timing of Start of systemIc Treatment for Asymptomatic Metastasized Pancreatic Cancer
Acronym: TIMEPAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.W. Wilmink, Dr. J.W. Wilmink, MD, PhD, Principal Investigator, Amsterdam UMC, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL722253.018.19
Record Dates: First submitted 2021-05-07; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate treatment (Active Comparator): The treatment schedule will be direct (start within 3 weeks of bate of diagnosis) FOLFIRINOX or nab paclitaxel in combination with gemcitabine per investigator's choice. Dosage and frequency of administration will be according to local protocol.
  Interventions: Drug: Folfirinox
- Delayed treatment (Active Comparator): The treatment schedule will be delayed treatment (based on symptoms) with FOLFIRINOX or nab paclitaxel in combination with gemcitabine per investigator's choice. Dosage and frequency of administration will be according to local protocol.
  Chemotherapy will start as soon as one of the following criteria is met:
  * Decline in performance status to ECOG < 1 or Karnofsky < 80%
  * Weight loss more than 5% of the total body weight from the time of study entry
  * Persistent nausea requiring medication
  * Pain requiring regular narcotic analgesics
  * Development of clinically significant third-space fluid collections
  * Liver function deterioration in the presence of progressive liver metastases
  Interventions: Drug: Folfirinox

INTERVENTIONS:
Drug: Folfirinox — In both arms the intervention will be FOLRINIOX or nab paclitaxel in combination with gemcitabine per investigator's choice

SUMMARY:
Since patients with metastatic pancreatic cancer have a limited life expectancy, it is important to determine the timing of when to start chemotherapy in order to optimize the benefits of chemotherapy relative to the side effects. Therefore, two treatment strategies can be considered: chemotherapy started immediately at diagnosis, or delayed until disease-related symptoms occur.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written Institutional Review Board/Ethics Committee-approved Informed Consent Form (ICF).
* Patients with histologically/cytological confirmed diagnosis of metastatic pancreatic ductal adenocarcinoma.
* Measurable disease on computed tomography (CT) scan per RECIST version 1.1 criteria.
* Eastern Cooperative Oncology Group Performance Status of 0-1
* Life expectancy ≥ 3 months.
* Age ≥ 18 years.
* A negative urine or serum pregnancy test within 7 days before Day 1 (first dose of study medication) if female subject is of childbearing potential.
* Screening clinical laboratory values as follows:

  1. Absolute neutrophil count > 1.5 x 109 /L
  2. Total bilirubin ≤ 1.5 times upper limit of normal (ULN).
  3. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times ULN, (if liver metastases are present, then ≤ 5 times ULN is allowed).
  4. Serum creatinine < 1.5 x ULN or creatinine clearance >50 mL/min/1.73 m2
  5. Prothrombin time/international normalized ratio within normal limits (± 15%) or within therapeutic range if subject takes warfarin. Partial thromboplastin time (PTT) within normal limits (± 15%).
  6. Platelet count > 100,000 x 109 /L
* No symptoms related to advanced disease, specified as:

  1. no pain requiring regular narcotic analgesics;
  2. no weight loss over 5 kg (unless related to surgery or other illness);
  3. no persistent nausea requiring medication;
  4. no obstructive bowel symptoms;
  5. no persistent fever related to metastatic cancer;
  6. no other symptom which in the opinion of the clinician was due to progressive metastatic cancer.
* No prior chemotherapy for metastatic disease (patients might have received adjuvant treatment more than 6 months before the development of metastatic disease, or neoadjuvant treatment before surgery for resectable disease)

Exclusion Criteria:

* Known central nervous system involvement or brain metastases.
* New York Heart Association Class III or IV cardiac disease or myocardial infarction within the past 12 months
* Any other disease, active, uncontrolled bacterial, viral or fungal infection requiring systemic therapy, metabolic dysfunction, physical examination finding or clinical laboratory finding that leads to reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or that may render the subject at high risk for treatment complications.
* Inability to comply with study and follow-up procedures as judged by the Investigator.
* Women currently pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-04-22 (Estimated); Study Completion 2024-04-22 (Estimated)

PRIMARY OUTCOMES:
Quality adjusted overall survival | From date of randomization until the date of death, assessed up to 12 months
  Measured in "utility-per-month", using the survival in months and the monthly reported quality of life by the EQ-5D-5L questionaire.

SECONDARY OUTCOMES:
Time to disease progression | 12 months
  Restricted mean progression free survival (RM-PFS): are under the Kaplan-Meier PFS curve between randomization and follow-up of the study (estimated 12 months)
Quality adjusted progression free survival (PFS) | From date of randomization until the date of death, assessed up to 12 months
Duration of time without symptoms of disease progression or toxicities (TWiST) | From date of randomization until the date of death, assessed up to 12 months
Overall survival | From date of randomization until the date of death, assessed up to 12 months
  (In months)
Number of patients with adverse events | From date of randomization until the date of death, assessed up to 12 months
  According to NCI CTC version 5.0

OTHER OUTCOMES:
Level of CA 19.9 | From date of randomization until the date of death, assessed up to 12 months
  Exploratory endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No